CLINICAL TRIAL: NCT05535738
Title: Biologics and Blistering - Using a Contact Dermatitis Model With Biologic Medications to Study Skin Inflammation Through Suction Blistering
Brief Title: Using a Contact Dermatitis Model With Biologic Medications to Study Skin Inflammation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wei-Che Ko (Other)
Responsible Party: Sponsor-Investigator, Wei-Che Ko, Professor of Dermatology, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000321
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-05

CONDITIONS: Skin Inflammation; Allergic Contact Dermatitis
Keywords: skin inflammation; allergic contact dermatitis
MeSH Terms: conditions — Dermatitis; Dermatitis, Allergic Contact | interventions — squaric acid dibutyl ester; dupilumab; Adalimumab; Ustekinumab; guselkumab; canakinumab; sarilumab; Triamcinolone Acetonide; Betamethasone Valerate; Fluticasone

STUDY DESIGN:
Intervention Model Description: There are two phases in this study. The first phase involves sensitization to a contact allergen and skin sampling to establish baseline characteristics. In the second phase, the participant will be pre-treated with a one time dose of an immunomodulating medication, re-treated with a contact allergen, followed by skin sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baseline Contact Allergen (Experimental): Individuals who will have allergic contact dermatitis induced via squaric acid dibutyl ester (SADBE) and/or known patch test allergens followed by skin and blood sampling. There is a protocol to sensitize individuals to SADBE if they have not previously been exposed to SADBE.
  Interventions: Drug: Squaric Acid Dibutyl Ester; Other: Known patch test allergens; Device: Microneedle; Device: Suction blistering; Procedure: Skin punch biopsy
- Contact Allergen with Immunomodulator Pre-Treatment (Experimental): Individuals from Arm 1 (Baseline Contact Allergen) who have been exposed to SADBE and/or known patch test allergens followed by skin and blood sampling. These individuals will be pre-treated via administration of a single dose of 1 biologic from the following list: dupilumab, adalimumab, ustekinumab, guselkumab, canakinumab, sarilumab; or a single application of 1 topical steroid from the following list: betamethasone valerate, triamcinolone acetonide, fluticasone propionate. Allergic contact dermatitis will then be induced and the skin sampled.
  Interventions: Drug: Squaric Acid Dibutyl Ester; Other: Known patch test allergens; Drug: Dupilumab; Drug: Adalimumab; Drug: Ustekinumab; Drug: Guselkumab; Drug: Canakinumab; Drug: Sarilumab; Drug: Triamcinolone Acetonide; Drug: Betamethasone Valerate; Drug: Fluticasone Propionate; Device: Microneedle; Device: Suction blistering; Procedure: Skin punch biopsy

INTERVENTIONS:
Drug: Squaric Acid Dibutyl Ester — Sensitization dose: 2% Elicitation doses: {0.0001%, 0.00025%, 0.00075%, 0.001%, 0.0025%, 0.005%, 0.0075%, 0.01%, 0.025%, 0.05%, 0.06%, 0.07%, 0.08%, 0.09%, 0.1%, 0.2%, 0.3%, 0.4%, 0.5%, 0.6% 0.7%, 0.8%, 0.9%, 1.0%, 1.2%, 1.4%, 1.6%, 1.8%, 2.0%}
Other: Known patch test allergens — Positive patch test allergens during the course of clinical patch testing will be re-applied on the back followed by skin sampling
Drug: Dupilumab — 300mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Adalimumab — 40mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Ustekinumab — 45mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Guselkumab — 100mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Canakinumab — 150mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Sarilumab — 200mg
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Triamcinolone Acetonide — 0.1% ointment
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Betamethasone Valerate — 0.1% ointment
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Drug: Fluticasone Propionate — 0.005% ointment
  Arms: Contact Allergen with Immunomodulator Pre-Treatment
Device: Microneedle — Painless and non-scarring skin sampling with a 7mm x 7mm patch of hydrogel-coated poly-l-lactide microneedles (<2mm length) will be used to collect interstitial fluid
Device: Suction blistering — Suction blistering is a technique to induce and collect blister fluid using a negative pressure instrument (Electronic Diversities Finksburg, MD). It does not require local anesthetic, stitches or pain medication following the procedure. The blisters will be no greater than 1cm in diameter and no deeper than the epidermis (<1mm deep). This process of inducing blisters is typically less than 1 hour. After the formation of blisters, the blister fluid will be extracted using a syringe. The blister roofs will be left attached to the skin and covered with petrolatum and a bandage.
Procedure: Skin punch biopsy — A skin biopsy is the removal of a small piece of tissue, under local anesthetic.

SUMMARY:
The purpose of this study is to answer: how do inflammation and anti-inflammatory skin therapies work in the skin? Inflammation is a protective response from the body's immune system to injury, disease, or irritation. It is a process by which your body's white blood cells and the things they make protect you from infection from outside invaders such as bacteria and viruses.

DETAILED DESCRIPTION:
The purpose of this study is to study mechanisms of human skin inflammation by using an established model of transient contact dermatitis with pre-treatment by biologic drugs that block specific inflammatory signals or by topical steroids that block broad inflammatory signals. Contact dermatitis will be induced in a safe and controlled manner through the use of topical application of squaric acid dibutyl ester (SADBE), along with other common allergens, after which skin will be sampled for analysis using nonscarring skin biopsy techniques including suction blister biopsies and/or application of absorptive microneedle patches.

This IRB protocol will use select FDA-approved, commercially available biologic drugs and topical steroids that have good safety profiles and block inflammatory signals that we observed in our previously acquired data of contact dermatitis.

This study will provide insight into human immunology that will deepen our understanding of dermatologic disease, as well as increase our understanding of topical steroids and biologic treatments which sometimes cause paradoxical inflammation despite being designed to suppress inflammation. We hope this will improve the basic understanding of human skin inflammation in order to ultimately impact treatment strategies for several skin diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects over the age of 18 years with no skin diseases
* Patients with dermatologic conditions such as atopic dermatitis, history of localized non-melanoma, keratinocytic skin cancer
* Patients with previous clinical patch testing
* UMass Medical School students and employees are eligible to participate.
* Non-English-speaking individuals are also eligible with the assistance of an interpreter and an approved short form consent in the appropriate language.

Exclusion Criteria:

* Adults unable to give consent
* History of the following specific dermatologic conditions (which would be confounders due to their particular immunologic etiologies, specifically the TNFa and IL-17 pathways which oppose the Th2 pathway): pityriasis rubra pilaris and psoriasis
* Patients actively receiving whole body phototherapy
* Patients actively receiving systemic broad-spectrum immunosuppression (prednisone, mycophenolate mofetil, azathioprine, methotrexate)
* Any history of poor wound healing
* History of uncontrolled diabetes
* History of easily torn skin
* Any known cardiac arrhythmia or history of heart failure
* History of demyelinating disease
* History of liver disease or alcohol abuse
* History of melanoma
* Pregnant women
* Individuals who are high risk for tuberculosis including prisoners, immigrants from TB- endemic areas, or US-based travelers who have visited TB-endemic areas
* Individuals with a self-reported personal history of infection with latent or active tuberculosis, HIV, Hepatitis B, or Hepatitis C will not be included, because the type of immunotherapies that will be used in this study may interfere with these conditions.
* For similar reasons, we will not be including individuals with signs of current or active infection, self-reported personal history of recurrent infections, or conditions that compromise the immune system, such as patients with malignancy (except non- melanoma, keratinocytic skin cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To collect and evaluate single-cell multiomics data (RNAseq, CITEseq, TCRseq) | Up to 5 years
  Baseline and after pre-treatment with immunomodulating medication

SECONDARY OUTCOMES:
Correlation of protein biomarkers collected by microneedles | Up to 5 years
  Correlation to RNA and/or protein expression collected by single-cell multiomics

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Che Ko, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States